CLINICAL TRIAL: NCT04068519
Title: Phase I/II Study Investigating Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activities of Anti-PD-1 Monoclonal Antibody BGB-A317 in Chinese Patients With Advanced Solid Tumors
Brief Title: Study Investigating Safety, Tolerability, Pharmacokinetics (PK) and Antitumor Activities of Anti-PD-1 (Programmed Death-1) Monoclonal Antibody
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-102
Record Dates: First submitted 2019-08-14; First posted 2019-08-28 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab (Experimental): Tislelizumab 200 mg intravenously (IV) once every 3 weeks (21 days per cycle) until no evidence of continued clinical benefits, unacceptable toxicity, or withdrawal of informed consent at the discretion of the investigator. There were 3 parts in this study: dose verification, pharmacokinetic (PK) sub-study, and indication expansion.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Administered intravenously
  Other Names: BGB-A317

SUMMARY:
This was a dose verification, pharmacokinetic (PK) assessment of products derived from two manufacturing processes and scales (500L-FMP and 2000L-FMP; FMP: Final Manufacturing Process) and indication expansion clinical study of monoclonal antibody conducted in Chinese subjects with advanced solid tumors, with a purpose of exploring the safety, tolerability, pharmacokinetics and preliminary efficacy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed advanced or metastatic tumors (unresectable), have had progression or intolerability since last standard anti-tumor treatment, or have no standard treatment or have refused standard therapy.
2. Participants must be able to provide archival tumor tissues (paraffin blocks or at least 10 unstained tumor specimen slides).
3. Participants must have at least one measurable lesion as defined per RECIST criterion version 1.1.
4. Participant must have adequate organ function.
5. Females are eligible to participate in the study if they are:

   a) Non-childbearing potential (that is, physiologically incapable of becoming pregnant) who:
   * Has had hysterectomy
   * Has had bilateral oophorectomy
   * Has had bilateral tubal ligation or are post-menopausal (total cessation of menses for ≥1 year) b) Childbearing potential:
   * Must be willing to use a highly effective method of birth control for the duration of the study, and for at least 120 days after the last dose of tislelizumab, and have a negative urine or serum pregnancy test within 7 days of the first dose of study drug.
6. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study.

Key Exclusion Criteria:

1. History of severe hypersensitivity reactions to other monoclonal antibodies (mAbs).
2. Prior malignancy active within the previous 2 years except for the tumor under investigation in this trial, cured or locally curable cancers, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.
3. Prior therapies targeting PD-1 or PD-L1. Active brain or leptomeningeal metastases. Participants with brain metastases are permitted if they are asymptomatic, for example, diagnosed incidentally by brain imaging, or participants with previously treated brain metastases that are asymptomatic at screening, radiographically stable and not requiring steroid medications for at least 4 weeks prior to the first administration of study treatment.
4. Participants with active autoimmune diseases or history of autoimmune diseases or immunodeficiency that may relapse should be excluded. Participants with following diseases are allowed to be enrolled for further screening: type I diabetes, hypothyroidism managed with hormone replacement therapy only, skin diseases not requiring systemic treatment (such as vitiligo, psoriasis or alopecia), or diseases not expected to recur in the absence of external triggering factors.
5. Participants should be excluded if they have a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of study drug administration.
6. With uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage.
7. Use of any live or attenuated vaccines within 4 weeks (28 days) prior to initiation of study therapy.
8. Major surgical procedure (Grade 3 or 4) within the past 4 weeks (28 days) prior to study drug administration.
9. Prior allogeneic or solid organ transplantation.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (12):
- China (12):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (North), Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital Sun Yat Sen University, Zhuhai, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Zhejiang University College of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Shen L, Guo J, Zhang Q, Pan H, Yuan Y, Bai Y, Liu T, Zhou Q, Zhao J, Shu Y, Huang X, Wang S, Wang J, Zhou A, Ye D, Sun T, Gao Y, Yang S, Wang Z, Li J, Wu YL. Tislelizumab in Chinese patients with advanced solid tumors: an open-label, non-comparative, phase 1/2 study. J Immunother Cancer. 2020 Jun;8(1):e000437. doi: 10.1136/jitc-2019-000437. PMID 32561638
- [Background] Zhou Q et al. Efficacy and safety data from a Phase 1/2 trial of tislelizumab in Chinese patients with non-small cell lung cancer. North America Conference on Lung Cancer, October 2020.
- [Derived] Ye D, Desai J, Shi J, Liu SM, Shen W, Liu T, Shi Y, Wang D, Liang L, Yang S, Ma X, Jin W, Zhang P, Huang R, Shen Z, Zhang Y, Wu YL. Co-enrichment of CD8-positive T cells and macrophages is associated with clinical benefit of tislelizumab in solid tumors. Biomark Res. 2023 Mar 7;11(1):25. doi: 10.1186/s40364-023-00465-w. PMID 36879284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 300 participants were treated with at least 1 dose of tislelizumab. This was a single arm study with 3 parts: dose verification, pharmacokinetic (PK) sub-study, and indication expansion.
Groups:
- Tislelizumab: Tislelizumab 200 mg was administered intravenously (IV) once every 3 weeks (21 days per cycle) until no evidence of continued clinical benefits, unacceptable toxicity, or withdrawal of informed consent at the discretion of the investigator.
Period: Dose Verification
Arm/Group | Tislelizumab
Started | 20
Completed | 4
Not Completed | 16
Not completed — Death | 15
Not completed — Withdrawal by Subject | 1
Period: Pharmacokinetic Sub-study
Arm/Group | Tislelizumab
Started | 57
Completed | 16
Not Completed | 41
Not completed — Death | 35
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 4
Not completed — Other not specified | 1
Period: Indication Expansion
Arm/Group | Tislelizumab
Started | 223
Completed | 54
Not Completed | 169
Not completed — Death | 152
Not completed — Withdrawal by Subject | 10
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) included all participants who received ≥ 1 dose of tislelizumab; Safety analysis data are summarized for the overall population given that the same dose was applied, regardless of part assignment, as pre-specified in the clinical study report.
Arm/Group | Tislelizumab
Number analyzed (Participants) | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 207
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 300

OUTCOME MEASURES:

1. Primary Outcome: Dose Verification and PK Sub-study: Number Participants With Adverse Events
Description: Number of participants with adverse events (AEs) and serious adverse events (SAEs), as defined per NCI-CTCAE Version 4.03, including physical examination, electrocardiograms and laboratory assessments
Time Frame: Up to approximately 23 months
Population: The Safety Analysis Set (SAS) included all participants who received ≥ 1 dose of tislelizumab
Measure: Count of Participants; unit: Participants
Groups:
- Dose Verification: Tislelizumab 200 mg intravenously (IV) once every 3 weeks (21 days per cycle) until no evidence of continued clinical benefits, unacceptable toxicity, or withdrawal of informed consent at the discretion of the investigator
- PK Sub-study: Tislelizumab 200 mg intravenously (IV) on Day 1 of the first 28 days followed by once every 3 weeks (21 days per cycle) for subsequent cycles until no evidence of continued clinical benefits, unacceptable toxicity, or withdrawal of informed consent at the discretion of the investigator
Arm/Group | Dose Verification | PK Sub-study
Number analyzed (Participants) | 20 | 57
Participants
  At least one treatment-emergent adverse event (TEAE) | 20 | 54
  TEAE Grade 3 of higher | 9 | 21
  Serious adverse event | 4 | 14

2. Primary Outcome: Dose Verification: Recommended Dose of Tislelizumab
Description: Recommended dose of tislelizumab for indication cohorts based on safety and tolerability
Time Frame: Up to approximately 23 months
Population: The Safety Analysis Set (SAS) included all participants who received ≥ 1 dose of tislelizumab
Measure: Number; unit: milligrams
Arm/Group | Dose Verification
Number analyzed (Participants) | 20
milligrams | 200

3. Primary Outcome: PK Sub-study: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of Tislelizumab From Two Manufacturing Processes and Scales
Description: Pharmacokinetics from products derived from two manufacturing scales at 500 liter and 2000 liter final manufacturing process (FMP) were evaluated
Time Frame: Predose, end of infusion, 3 hours, 6 hours on Day 1, Day 2, Day 4, Day 8, Day 15, Day 22, and Day 29 predose
Population: The PK Analysis Set included participants in the SAS for whom at least 1 valid PK parameter could be derived for tislelizumab
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL*day
Arm/Group | PK Sub-study
Number analyzed (Participants) | 56
µg/mL*day
  500L-FMP: number analyzed (Participants) | 25
  500L-FMP | 1113.9 [997.6 to 1244]
  2000L-FMP: number analyzed (Participants) | 31
  2000L-FMP | 1108 [985.2 to 1246]

4. Primary Outcome: PK Sub-study: Area Under the Concentration-time Curve From Time 0 to 28 Days Postdose (AUC0-28d) of Tislelizumab From Two Manufacturing Processes and Scales
Description: as for outcome 3
Time Frame: Predose, end of infusion, 3 hours, 6 hours on Day 1, Day 2, Day 4, Day 8, Day 15, Day 22, and Day 29 predose
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL*day
Arm/Group | PK Sub-study
Number analyzed (Participants) | 56
µg/mL*day
  500L-FMP: number analyzed (Participants) | 25
  500L-FMP | 810.2 [746.0 to 879.9]
  2000L-FMP: number analyzed (Participants) | 31
  2000L-FMP | 801.7 [740.8 to 867.5]

5. Primary Outcome: PK Sub-study: Maximum Observed Concentration (Cmax) of Tislelizumab From Two Manufacturing Processes and Scales
Description: Pharmacokinetics from products derived from two manufacturing scales at 500 liter and 2000 liter FMP were evaluated
Time Frame: Predose, end of infusion, 3 hours, 6 hours on Day 1, Day 2, Day 4, Day 8, Day 15, Day 22, and Day 29 predose
Population: PK Analysis Set included participants in the SAS for whom at least 1 valid PK parameter could be derived for tislelizumab
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | PK Sub-study
Number analyzed (Participants) | 56
µg/mL
  500L-FMP: number analyzed (Participants) | 25
  500L-FMP | 77.3 [73.6 to 81.2]
  2000L-FMP: number analyzed (Participants) | 31
  2000L-FMP | 75.7 [70.7 to 81.0]

6. Primary Outcome: Indication Expansion: Objective Response Rate
Description: Objective response rate (ORR) is defined as the percentage of participants who achieved objective tumor response (complete response or partial response) according to RECIST Version 1.1. Indication expansion includes participants from all parts in the following indications: non-small cell lung cancer (NSCLC), melanoma, esophageal squamous cell carcinoma (ESCC), gastric cancer (GC), urothelial carcinoma (UC), nasopharyngeal carcinoma (NPC), renal cell carcinoma (RCC), hepatocellular carcinoma (HCC), microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) tumors, and other tumor types.
Time Frame: Up to approximately 3 years and 5 months
Population: The Safety Analysis Set (SAS) included all participants who received ≥ 1 dose of tislelizumab; one participant is included in both MSI-H/dMMR and GC indications.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 300
Percentage of participants
  NSCLC: number analyzed (Participants) | 56
  NSCLC | 17.9 [8.9 to 30.4]
  Melanoma: number analyzed (Participants) | 34
  Melanoma | 17.6 [6.8 to 34.5]
  ESCC: number analyzed (Participants) | 26
  ESCC | 7.7 [0.9 to 25.1]
  GC: number analyzed (Participants) | 24
  GC | 16.7 [4.7 to 37.4]
  UC: number analyzed (Participants) | 22
  UC | 18.2 [5.2 to 40.3]
  NPC: number analyzed (Participants) | 21
  NPC | 47.6 [25.7 to 70.2]
  RCC: number analyzed (Participants) | 21
  RCC | 9.5 [1.2 to 30.4]
  HCC: number analyzed (Participants) | 18
  HCC | 16.7 [3.6 to 41.4]
  MSI-H/dMMR: number analyzed (Participants) | 16
  MSI-H/dMMR | 25.0 [7.3 to 52.4]
  Other: number analyzed (Participants) | 63
  Other | 9.5 [3.6 to 19.6]

7. Secondary Outcome: Dose Verification: Area Under the Concentration-time Curve From Time 0 to 21 Days Postdose (AUC0-tau) of Tislelizumab
Time Frame: Predose, end of infusion, 1.5 hours, 6 hours on Day 1, Day 2, Day 4, Day 8, Day 15, Day 22 predose in Cycle 1 and Cycle 5 (21 days per cycle)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µg/mL*day
Arm/Group | Dose Verification
Number analyzed (Participants) | 20
µg/mL*day
  Cycle 1 | 600.1 (144.5)
  Cycle 5: number analyzed (Participants) | 12
  Cycle 5 | 1122 (352)

8. Secondary Outcome: Dose Verification: Maximum Observed Concentration (Cmax) of Tislelizumab
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Dose Verification
Number analyzed (Participants) | 20
µg/mL
  Cycle 1 | 67.8 (12.8)
  Cycle 5: number analyzed (Participants) | 12
  Cycle 5 | 131 (37.7)

9. Secondary Outcome: Dose Verification: Predose Plasma Concentration of Tislelizumab During Multiple Dosing (Ctrough)
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Dose Verification
Number analyzed (Participants) | 15
µg/mL
  Cycle 1 | 15.8 (4.73)
  Cycle 5: number analyzed (Participants) | 11
  Cycle 5 | 31.4 (9.55)

10. Secondary Outcome: Dose Verification: Apparent Terminal Half-life of Tislelizumab (t1/2)
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dose Verification
Number analyzed (Participants) | 19
Days
  Cycle 1 | 13.3 (2.95)
  Cycle 5: number analyzed (Participants) | 10
  Cycle 5 | 16.9 (3.79)

11. Secondary Outcome: Dose Verification: Clearance (Cl)
Time Frame: Predose, end of infusion, 1.5 hours, 6 hours on Day 1, Day 2, Day 4, Day 8, Day 15, Day 22 predose in Cycle 1 (21 days per cycle)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | Dose Verification
Number analyzed (Participants) | 20
Liters/day | 0.247 (0.0918)

12. Secondary Outcome: Indication Expansion: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from the date of first study dose to disease progression or death, whichever comes first, as determined by Investigator per RECIST version 1.1. Indication expansion includes participants from all parts in the following indications: non-small cell lung cancer (NSCLC), melanoma, esophageal squamous cell carcinoma (ESCC), gastric cancer (GC), urothelial carcinoma (UC), nasopharyngeal carcinoma (NPC), renal cell carcinoma (RCC), hepatocellular carcinoma (HCC), microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) tumors, and other tumor types.
Time Frame: Up to approximately 3 years and 5 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Tislelizumab: Tislelizumab 200 mg intravenously (IV) once every 3 weeks (21 days per cycle) until no evidence of continued clinical benefits, unacceptable toxicity, or withdrawal of informed consent at the discretion of the investigator.
Arm/Group | Tislelizumab
Number analyzed (Participants) | 300
Months
  NSCLC: number analyzed (Participants) | 56
  NSCLC | 4.0 [2.1 to 8.1]
  Melanoma: number analyzed (Participants) | 34
  Melanoma | 2.2 [2.0 to 6.1]
  ESCC: number analyzed (Participants) | 26
  ESCC | 2.1 [2.0 to 4.2]
  GC: number analyzed (Participants) | 24
  GC | 2.1 [1.9 to 4.0]
  UC: number analyzed (Participants) | 22
  UC | 2.1 [2.0 to 4.3]
  NPC: number analyzed (Participants) | 21
  NPC | 8.2 [4.2 to 11.4]
  RCC: number analyzed (Participants) | 21
  RCC | 4.1 [2.1 to 10.4]
  HCC: number analyzed (Participants) | 18
  HCC | 4.0 [2.1 to 12.4]
  MSI-H/dMMR: number analyzed (Participants) | 16
  MSI-H/dMMR | 6.1 [2.0 to 15.3]
  Other: number analyzed (Participants) | 63
  Other | 2.3 [2.2 to 2.8]

13. Secondary Outcome: Indication Expansion: Duration of Response
Description: Duration of response for responders with complete or partial response is defined as the time interval between the date of the earliest qualifying response and the date of progressive disease or death for any cause, whichever occurs earlier as determined by Investigator per RECIST version 1.1. Indication expansion includes participants from all parts in the following indications: non-small cell lung cancer (NSCLC), melanoma, esophageal squamous cell carcinoma (ESCC), gastric cancer (GC), urothelial carcinoma (UC), nasopharyngeal carcinoma (NPC), renal cell carcinoma (RCC), hepatocellular carcinoma (HCC), microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) tumors, and other tumor types.
Time Frame: Up to approximately 3 years and 5 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 51
Months
  NSCLC: number analyzed (Participants) | 10
  NSCLC | 30.4 [8.3 to 30.4]
  Melanoma: number analyzed (Participants) | 6
  Melanoma | 12.5 [4.2 to NA] — Not estimable due to insufficient number of participants with events
  ESCC: number analyzed (Participants) | 2
  ESCC | NA [13.8 to NA] — Not estimable due to insufficient number of participants with events
  GC: number analyzed (Participants) | 4
  GC | NA [13.9 to NA] — Not estimable due to insufficient number of participants with events
  UC: number analyzed (Participants) | 4
  UC | NA [8.3 to NA] — Not estimable due to insufficient number of participants with events
  NPC: number analyzed (Participants) | 10
  NPC | 8.8 [3.9 to 14.8]
  RCC: number analyzed (Participants) | 2
  RCC | NA [4.4 to NA] — Not estimable due to insufficient number of participants with events
  HCC: number analyzed (Participants) | 3
  HCC | NA [8.3 to NA] — Not estimable due to insufficient number of participants with events
  MSI-H/dMMR: number analyzed (Participants) | 4
  MSI-H/dMMR | NA [5.1 to NA] — Not estimable due to insufficient number of participants with events
  Other: number analyzed (Participants) | 6
  Other | NA [8.3 to NA] — Not estimable due to insufficient number of participants with events

14. Secondary Outcome: Indication Expansion: Clinical Benefit Rate
Description: Clinical benefit rate is defined as the percentage of participants in specific tumor types reaching confirmed CR, PR and durable stable disease (SD; at ≥ 24 weeks) in accordance with RECIST version 1.1. Indication expansion includes participants from all parts in the following indications: non-small cell lung cancer (NSCLC), melanoma, esophageal squamous cell carcinoma (ESCC), gastric cancer (GC), urothelial carcinoma (UC), nasopharyngeal carcinoma (NPC), renal cell carcinoma (RCC), hepatocellular carcinoma (HCC), microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) tumors, and other tumor types.
Time Frame: Up to approximately 3 years and 5 months
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 300
Percentage of participants
  NSCLC: number analyzed (Participants) | 56
  NSCLC | 33.9 [21.8 to 47.8]
  Melanoma: number analyzed (Participants) | 34
  Melanoma | 32.4 [17.4 to 50.5]
  ESCC: number analyzed (Participants) | 26
  ESCC | 15.4 [4.4 to 34.9]
  GC: number analyzed (Participants) | 24
  GC | 25.0 [9.8 to 46.7]
  UC: number analyzed (Participants) | 22
  UC | 27.3 [10.7 to 50.2]
  NPC: number analyzed (Participants) | 21
  NPC | 61.9 [38.4 to 81.9]
  RCC: number analyzed (Participants) | 21
  RCC | 38.1 [18.1 to 61.6]
  HCC: number analyzed (Participants) | 18
  HCC | 38.9 [17.3 to 64.3]
  MSI-H/dMMR: number analyzed (Participants) | 16
  MSI-H/dMMR | 50.0 [24.7 to 75.3]
  Other: number analyzed (Participants) | 63
  Other | 22.2 [12.7 to 34.5]

15. Secondary Outcome: Indication Expansion: Overall Survival
Description: Overall survival is defined as the time from the date of the first study dose to death. Indication expansion includes participants from all parts in the following indications: non-small cell lung cancer (NSCLC), melanoma, esophageal squamous cell carcinoma (ESCC), gastric cancer (GC), urothelial carcinoma (UC), nasopharyngeal carcinoma (NPC), renal cell carcinoma (RCC), hepatocellular carcinoma (HCC), microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) tumors, and other tumor types.
Time Frame: Up to approximately 3 years and 5 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab
Number analyzed (Participants) | 300
Months
  NSCLC: number analyzed (Participants) | 56
  NSCLC | 22.1 [10.1 to 33.5]
  Melanoma: number analyzed (Participants) | 34
  Melanoma | 11.8 [7.0 to 24.2]
  ESCC: number analyzed (Participants) | 26
  ESCC | 4.8 [3.6 to 8.5]
  GC: number analyzed (Participants) | 24
  GC | 4.7 [2.4 to 14.6]
  UC: number analyzed (Participants) | 22
  UC | 4.3 [2.1 to 22.9]
  NPC: number analyzed (Participants) | 21
  NPC | 25.0 [11.7 to NA] — Not estimable due to insufficient number of participants with events
  RCC: number analyzed (Participants) | 21
  RCC | 19.8 [8.0 to 24.3]
  HCC: number analyzed (Participants) | 18
  HCC | 25.1 [5.5 to NA] — Not estimable due to insufficient number of participants with events
  MSI-H/dMMR: number analyzed (Participants) | 16
  MSI-H/dMMR | 19.4 [4.2 to NA] — Not estimable due to insufficient number of participants with events
  Other: number analyzed (Participants) | 63
  Other | 9.0 [4.8 to 13.4]

16. Secondary Outcome: Indication Expansion: Disease Control Rate
Description: Disease control rate is defined as the percentage of participants reaching CR, PR, and SD according to RECIST version 1.1. Indication expansion includes participants from all parts in the following indications: non-small cell lung cancer (NSCLC), melanoma, esophageal squamous cell carcinoma (ESCC), gastric cancer (GC), urothelial carcinoma (UC), nasopharyngeal carcinoma (NPC), renal cell carcinoma (RCC), hepatocellular carcinoma (HCC), microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) tumors, and other tumor types.
Time Frame: Up to approximately 3 years and 5 months
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 300
Percentage of participants
  NSCLC: number analyzed (Participants) | 56
  NSCLC | 55.4 [41.5 to 68.7]
  Melanoma: number analyzed (Participants) | 34
  Melanoma | 38.2 [22.2 to 56.4]
  ESCC: number analyzed (Participants) | 26
  ESCC | 34.6 [17.2 to 55.7]
  GC: number analyzed (Participants) | 24
  GC | 25.0 [9.8 to 46.7]
  UC: number analyzed (Participants) | 22
  UC | 40.9 [20.7 to 63.6]
  NPC: number analyzed (Participants) | 21
  NPC | 81.0 [58.1 to 94.6]
  RCC: number analyzed (Participants) | 21
  RCC | 52.4 [29.8 to 74.3]
  HCC: number analyzed (Participants) | 18
  HCC | 55.6 [30.8 to 78.5]
  MSI-H/dMMR: number analyzed (Participants) | 16
  MSI-H/dMMR | 50.0 [24.7 to 75.3]
  Other: number analyzed (Participants) | 63
  Other | 31.7 [20.6 to 44.7]

17. Secondary Outcome: Number of Participants With Positive Anti-drug Antibody (ADA) Status to Tislelizumab
Time Frame: Up to approximately 23 months
Population: Evaluable participants had non-missing baseline ADA and at least 1 non-missing postbaseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Tislelizumab
Number analyzed (Participants) | 279
Participants
  Treatment-emergent | 43
  Treatment-boosted | 2
  Treatment-induced | 41

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study treatment; Up to approximately 3 years and 5 months
Description: All AEs will be recorded during the study (AE from the time of the first dose and SAEs from the time of signing of informed consent) and for up to 30 days after the last dose of study treatment or until the initiation of another anticancer therapy, whichever occurs first.
Groups:
- Tislelizumab: Tislelizumab 200 mg was administered intravenously (IV) once every 3 weeks (21 days per cycle) until no evidence of continued clinical benefits, unacceptable toxicity, or withdrawal of informed consent at the discretion of the investigator. Safety analysis data are summarized for the overall population given that the same dose was applied, regardless of part assignment, as pre-specified in the clinical study report.
Arm/Group | Tislelizumab
All-Cause Mortality (participants affected / at risk) | 202/300
Serious Adverse Events (participants affected / at risk) | 85/300
Other Adverse Events (participants affected / at risk) | 277/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab (N=300)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Immune-mediated myocarditis (Cardiac disorders) | 2 (3)
Cataract (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 4 (4)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (8)
Vomiting (Gastrointestinal disorders) | 2 (4)
Death (General disorders) | 5 (5)
Fatigue (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (6)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 11 (13)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Anastomotic fistula (Injury, poisoning and procedural complications) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Blood magnesium decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Brain oedema (Nervous system disorders) | 1 (2)
Cerebral artery embolism (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Lacunar infarction (Nervous system disorders) | 1 (1)
Paralysis (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab (N=300)
Anaemia (Blood and lymphatic system disorders) | 110 (227)
Leukopenia (Blood and lymphatic system disorders) | 9 (22)
Hyperthyroidism (Endocrine disorders) | 14 (15)
Hypothyroidism (Endocrine disorders) | 45 (67)
Abdominal pain (Gastrointestinal disorders) | 11 (14)
Constipation (Gastrointestinal disorders) | 29 (37)
Diarrhoea (Gastrointestinal disorders) | 21 (25)
Dysphagia (Gastrointestinal disorders) | 9 (13)
Nausea (Gastrointestinal disorders) | 19 (24)
Vomiting (Gastrointestinal disorders) | 19 (23)
Fatigue (General disorders) | 20 (22)
Malaise (General disorders) | 26 (32)
Non-cardiac chest pain (General disorders) | 12 (13)
Pyrexia (General disorders) | 39 (63)
Pneumonia (Infections and infestations) | 11 (21)
Upper respiratory tract infection (Infections and infestations) | 26 (33)
Urinary tract infection (Infections and infestations) | 11 (14)
Alanine aminotransferase increased (Investigations) | 71 (129)
Aspartate aminotransferase increased (Investigations) | 81 (138)
Bilirubin conjugated increased (Investigations) | 37 (127)
Blood albumin decreased (Investigations) | 9 (13)
Blood alkaline phosphatase increased (Investigations) | 24 (40)
Blood bilirubin increased (Investigations) | 52 (186)
Blood bilirubin unconjugated increased (Investigations) | 21 (87)
Blood creatine phosphokinase increased (Investigations) | 16 (38)
Blood creatinine increased (Investigations) | 16 (37)
Blood glucose increased (Investigations) | 13 (28)
Blood lactate dehydrogenase increased (Investigations) | 22 (33)
Blood thyroid stimulating hormone increased (Investigations) | 13 (14)
Blood triglycerides increased (Investigations) | 13 (36)
Blood urea increased (Investigations) | 12 (40)
Blood uric acid increased (Investigations) | 14 (35)
Gamma-glutamyltransferase increased (Investigations) | 47 (102)
Haemoglobin decreased (Investigations) | 12 (20)
Neutrophil count decreased (Investigations) | 22 (80)
Neutrophil count increased (Investigations) | 14 (14)
Platelet count decreased (Investigations) | 26 (74)
Protein urine present (Investigations) | 17 (22)
Red blood cells urine positive (Investigations) | 17 (34)
Weight decreased (Investigations) | 50 (82)
Weight increased (Investigations) | 33 (97)
White blood cell count decreased (Investigations) | 36 (137)
White blood cells urine positive (Investigations) | 19 (34)
Decreased appetite (Metabolism and nutrition disorders) | 27 (29)
Hyperglycaemia (Metabolism and nutrition disorders) | 17 (28)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 12 (34)
Hyperuricaemia (Metabolism and nutrition disorders) | 22 (55)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 34 (64)
Hypokalaemia (Metabolism and nutrition disorders) | 21 (38)
Hyponatraemia (Metabolism and nutrition disorders) | 21 (45)
Hypophosphataemia (Metabolism and nutrition disorders) | 10 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (23)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (14)
Dizziness (Nervous system disorders) | 11 (14)
Insomnia (Psychiatric disorders) | 18 (18)
Proteinuria (Renal and urinary disorders) | 52 (114)
Cough (Respiratory, thoracic and mediastinal disorders) | 36 (48)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 (18)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 16 (27)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (30)
Rash (Skin and subcutaneous tissue disorders) | 25 (45)
Hypertension (Vascular disorders) | 14 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT04068519/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT04068519/SAP_001.pdf